CLINICAL TRIAL: NCT02531256
Title: An Investigation of a New Laryngeal Mask Airway LMA Protector
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013/709/D
Record Dates: First submitted 2015-08-21; First posted 2015-08-24 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2015-08

CONDITIONS: Airway Morbidity
Keywords: Laryngeal Mask Airway

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LMA Protector (Experimental): Single Use Supraglottic Airway Device with 2 ports for gastric access (male and female port)
  Interventions: Device: LMA Protector

INTERVENTIONS:
Device: LMA Protector — Insertion of airway device for airway management during gynaecological procedure

SUMMARY:
Evaluation of LMA Protector

DETAILED DESCRIPTION:
This new disposable silicone airway device provides access and functional separation of the respiratory and digestive tracts. The airway tube is elliptical in cross section ending at the laryngeal opening. The device contains 2 drainage channels (male and female port) proximally that continues into a common distal opening posterior to the distal airway cuff bowl. The female port allows a gastric tube to be passed into the stomach, whilst a suction tube may be attached to the male suction port offering removal of gastric fluid around the upper oesophagus sphincter.

ELIGIBILITY:
Inclusion Criteria:

* planned elective surgery with indication for LMA use

Exclusion Criteria:

* body mass index of 30 or more, known gastro-oesophageal reflux, patients with increased risk of aspiration, upper airway pathology and mouth opening of less than 2 cm

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of insertion attempts | 5 minutes
  Time of pickup of device to the presence of carbon dioxide trace on

SECONDARY OUTCOMES:
Oropharyngeal Leak Pressure | 5 minutes
  Closure of expiratory valve of circle anaesthetic breathing system and noting the airway pressure in the breathing system at equilibration with cuff pressure of 60cmH2O or up to maximum of 40cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Ban L Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sng BL, Ithnin FB, Mathur D, Lew E, Han NR, Sia AT. A preliminary assessment of the LMA protector in non-paralysed patients. BMC Anesthesiol. 2017 Feb 20;17(1):26. doi: 10.1186/s12871-017-0323-5. PMID 28219323